CLINICAL TRIAL: NCT05824325
Title: Different Targeted Antibody-drug Conjugates for HER2 Ultra-low or no Expression Advanced Breast Cancer: a Phase Ⅰb/Ⅱ Study（GALAXY）
Brief Title: Different Targeted Antibody-drug Conjugates For HER2 Ultra-low or No Expression Advanced Breast Cancer（GALAXY）
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Chief Physician, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GALAXY
Record Dates: First submitted 2023-03-05; First posted 2023-04-21 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: HER2 ADC (Experimental): Patients diagnosed with HER2 ultra-low or no expression are recruited
  Interventions: Drug: SHR-A1811
- Experimental: TROP2 ADC (Experimental): Patients diagnosed with HER2 ultra-low or no expression are recruited.
  Interventions: Drug: TROP2 ADC

INTERVENTIONS:
Drug: SHR-A1811 — HER2 ADC
  Arms: Experimental: HER2 ADC
Drug: TROP2 ADC — TROP2 ADC
  Arms: Experimental: TROP2 ADC

SUMMARY:
This is a phaseⅠb/Ⅱ, open-label, two-arm parallel study evaluating the efficacy and safety of different targeted antibody-drug conjugates for HER2 ultra-low or no expression advanced breast cancer

ELIGIBILITY:
Inclusion Criteria:

ECOG Performance Status of 0 or 1

Pathologically documented breast cancer that:

1. is advanced or metastatic
2. is histologically confirmed to be HER2 IHC 0 (ISH- or untested)
3. was never previously HER2-positive (IHC 3+ or ISH+) At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.

Disease progression on at least 1 previous line of chemotherapy for recurrent/metastatic breast cancer. Subjects with HER2-negative and hormone-receptor positive tumors must have progressed after at least 1 line of endocrine therapy with or without CDK4/6 inhibitor.

Has protocol-defined adequate organ and bone marrow function. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

Has previously been treated with any anti-HER2 therapy. Known prior severe hypersensitivity to investigational product or any component in its formulation and other monoclonal antibodies.

Any major surgery, radiotherapy, chemotherapy, immunotherapy or molecular targeted therapy, biotherapy or other drug clinical trial within 4 weeks; received endocrine therapy within 2 weeks before the first study drug administration.

History of other malignancy than breast cancer within 5 years prior to screening (except for cured skin basal cell carcinoma and cervical carcinoma in situ).

Meningeal metastasis or active brain parenchymal metastasis. Any concurrent use of immunosuppressant or systemic corticosteroid treatment to achieve immunosuppression purpose (dose of > 10mg/day prednisone or equivalent), and still in use within 2 weeks before the first study drug administration.

Has uncontrolled intercurrent illness or significant cardiovascular disease. History of clinically significant lung diseases. History of immunodeficiency, including HIV positive. Known active hepatitis B virus or hepatitis C virus infection. Has any medical history or condition that per protocol or in the opinion of the investigator is inappropriate for the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 56 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-04-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events (AEs)- Phase 1 | Up to follow-up period, approximately 24 months
  Occurrence of AEs in Phase 1 graded according to CTCAE v5.0
Objective Response Rate (ORR)- Phase 2 | Until progression, assessed up to approximately 24 months
  The proportion of patients who have a CR or PR, as determined by the Investigator at local site per RECIST 1.1.

SECONDARY OUTCOMES:
Progression Free Survival (PFS | Until progression, assessed up to approximately 24 months
  Time to progression as assessed by the Investigator at local site per RECIST 1.1, or death due to any cause.
Overall Survival (OS) | Until death, assessed up to approximately 24 months
  time to death due to any cause
Duration of Response (DoR) | Until progression, assessed up to approximately 24 months
  Time from the date of first documented response until the date of documented progression or death in the absence of disease progression.
Disease Control Rate (DCR) | Baseline through end of study, assessed up to 24 months
  The proportion of patients who have a CR or PR or SD, as determined by the Investigator at local site per RECIST 1.1.
Clinical Benefit Rate (CBR) | Until progression or death, assessed up to approximately 24 months
  The percentage of subjects with CR, PR and SD≥24 weeks，as determined by the Investigator at local site per RECIST 1.1.
Exploratory analyses | Baseline until disease progression or loss of clinical benefit, assessed up to 24 months
  HER2-PET was done at baseline to further explore the clinical utility of HER2-PET for HER2 detection
Safety | Up to follow-up period, approximately 24 months
  Occurrence of Adverse Events(AEs) graded according to CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China